CLINICAL TRIAL: NCT02575287
Title: Mucosal and Minimal Injuries Detected Through Digital Chromoendoscopy Using Optical Enhancement System™ Associated to High Definition Plus Optical Magnification in Non Erosive Gastroesophageal Reflux Disease
Brief Title: Minimal Injuries From Esophagus Detected by Optical Enhancement System™ Associated to Optical Magnification HD Scopes
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: I-JUN-17-2015
Record Dates: First submitted 2015-09-09; First posted 2015-10-14 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Non Erosive Reflux Disease; GERD
MeSH Terms: conditions — Non-Erosive Reflux Disease; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — histological biopsies from esophagus
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NERD group: (Digital chromoendoscopy with Optical Enhancement and without magnification; Digital chromoendoscopy with Optical Enhancement and with magnification; optical magnification without Digital chromoendoscopy: Optical Enhancement) Patients with reflux symptoms, without endoscopic lesions on the upper endoscopy with high definition white light or I-Scan and a positive ph-impedanciometry for reflux
  Interventions: Device: Optical Enhancement; Device: Optical Enhancement with optical magnification; Device: Optical magnification without Optical enhancement
- Control group: (Digital chromoendoscopy with Optical Enhancement and without magnification; Digital chromoendoscopy with Optical Enhancement and with magnification; optical magnification without Digital chromoendoscopy: Optical Enhancement) Patients with reflux symptoms, without endoscopic lesions on the upper endoscopy with high definition white light or I-Scan and a negative ph-impedanciometry for reflux
  Interventions: Device: Optical Enhancement; Device: Optical Enhancement with optical magnification; Device: Optical magnification without Optical enhancement

INTERVENTIONS:
Device: Optical Enhancement — A endoscopic visualization of the mucosa using the pre-processor filter called Optical enhancement (Pentax Video Processor EPK-i7010; HOYA Co. Tokyo, Japan)
  Other Names: OE system
Device: Optical Enhancement with optical magnification — A endoscopic visualization of the mucosa using the pre-processor filter called Optical enhancement associated with an optical magnification using the scope called magniview (PENTAX Medical EG-2990Zi)
  Other Names: OE sytem with optical magnification
Device: Optical magnification without Optical enhancement — A endoscopic visualization of the mucosa using optical magnification without the use of the pre-processor filter called Optical enhancement
  Other Names: Optical magnification without OE sytem

SUMMARY:
White light endoscopy remains the gold standard technique to evaluate gastrointestinal tract. Gastroesophageal Reflux Disease (GERD) is defined as presence of reflux symptoms (heartburn and regurgitation) associated or not with lesions in esophageal mucosa. Based on findings at videoendoscopy GERD patients can have a complicated reflux disease (erosive esophagitis) or not and be considered as a non erosive reflux disease (NERD). 60% of GERD patients have normal endoscopy (NERD) and requires further studies to achieve a definitive diagnosis. Based on this fact is that the study will be focus on NERD patients.

Recently an image-enhanced endoscopic technology using a pre-processor band-limited light called Optical Enhancement system (OE system™), was developed (Pentax Medical). This new technology combines digital signal processing with optical filters that limit the spectral characteristics of the illumination light. The new innovated optical filters achieve higher overall transmittance by connecting the peaks of the hemoglobin absorption spectrum (415 nm, 540 nm and 570 nm) creating a continuous wavelength spectrum. There are two modes with different OE filters (Mode 1 and Mode 2). Mode 1 is designed to improve visualization of microvessels with a sufficient amount of light, and Mode 2 is designed to improve contrast of white-light observation by bringing the color tone of the overall image closer to that of natural color.

In addition, new scopes has been developed which combines high definition images with optical magnification called Magniview™. These scopes increase the image up to 136 times with a better quality of image than standard scopes without optical zoom. Sharma et al. evaluated esophageal changes in NERD patients using a similar pre-processor filter called Narrow Band Imaging (NBI). They found that a significantly higher proportion of patients with NERD had an increased number, dilation and tortuosity of the microscopic intrapapillary capillary loops (IPCLs), and were considered the best predictors for diagnosing NERD. They used optical chromoendoscopy technology (NBI) associated to magnification scopes (Olympus GIF Q240Z, 115x), but they did not evaluated if the contribution with this technology to the observations found in GERD patients were as a result of the NBI or the magnification scopes. The investigators opinion is that chromoendoscopy is useful but is the magnification what makes up the difference.

DETAILED DESCRIPTION:
Sharma et al. described in detail the changes of the intrapapillary capillaries seen with reflux inflammation. In the normal esophageal mucosa, submucosa all vessels are connected to the arborescent vascular network. Intrapapillary capillaries arise from the fourth branch of the arborescent vessels into the epithelial papillae and form single loops called IPCLs. It has been shown that IPCLs dilate and elongate along with an increase in the number and density of arborescent vessels in mucosal cancer. These changes are similar to those observed in inflammation.

Estimated enrollment: 100 patients (NERD group: 50 patients and control group: 50 patients)

Study design: This is an observational and analytical cross-section, population - based survey study, with prospective case collection, non-randomized and simple blind, performed in a Tertiary Academic Center.

Study Design

* Allocation: Non randomized, simple blind
* Endpoint Classification: Efficacy
* Intervention Model: Non interventional
* Primary Purpose: Diagnosis

Setting: Instituto Ecuatoriano de Enfermedades Digestivas (IECED), OmniHospital Academic Tertiary Center. We will include patients from September 2015 to November 2015. Patients will be recruited from the gastroenterology unit (IECED). The study protocol and consent form has been approved by the IRB and will be conducted according to the declaration of Helsinki. Patients will sign an informed consent and answer a questionnaire that includes constitutional data (sex, age, weight (Kg), height (m), BMI (Kg/m2), chronic diseases, medication and main reflux symptom).

Population selection, inclusion and exclusion criteria: Patient selection was done after the following analysis. Each patients that had reflux symptoms (heartburn and regurgitation) and 8 or more points at the Spanish version of GERD questionnaire validated by Zavala-González et al., underwent an upper videoendoscopy using initially high definition white light and then virtual chromoendoscopy (I-Scan™) in the three different image algorithms. After performing an upper endoscopy completely and reach the line Z, the entire esophagus was evaluated (upper, middle and lower esophagus). If they had any signs of reflux as ulcerative esophagitis, esophageal strictures, Barrett's esophagus or any erosive sign according to Los Angeles classification (Grade A to D), they were classified as GERD patients and were excluded from the protocol. The endoscopies were performed by the same three endoscopist that will carry on the study.

If the esophagus was normal and no changes were seen by these two techniques, they were considered as NERD patients and a pH-impedanciometry was performed as gold standard study, in order to diagnosis reflux disease. GERD diagnosis was considered when there were more than 73 episodes of reflux episodes in 24 hours or acid exposure time (AET) abnormal with ph <4 measured in more than 4,2%of the time over 24 hours.

After this phase, the investigators could discriminate patients that had a normal pH-impedanciometry and no reflux disease from the real NERD patients with reflux disease proven by a positive pH-impedanciometry with symptoms and no lesion.

Two groups were selected. One was the control group and included patients that agreed to be part of the study and for whom we have certainty that they have no GERD (reflux symptoms but negative upper endoscopy with high definition white light or I-Scan and negative Ph-impedanciometry). The other group includes NERD patients with reflux symptoms, a positive Ph-Impedanciometry but a negative upper endoscopy with high definition white light or I-Scan.

Survey: It will be use the Spanish version of the Gastroesophageal Reflux Disease Questionnaire survey, validated in Mexico by Zavala-González et al., but in an Ecuadorian population.

1. How often did you have a burning feeling behind your breastbone (heartburn)?
2. How often did you have stomach contents (liquid or food) moving upwards to your throat or mouth (regurgitation)?
3. How often did you have pain in the center of the upper stomach?
4. How often did you have nausea?
5. How often did you have difficulty getting a good night's sleep because of your heartburn and/or regurgitation?
6. How often did you take additional medication for your heartburn and/or regurgitation, other than what the physician told you to take (such as Tums, Rolaids and Maalox)?

Endoscopic technique: All the patients included in the protocol (NERD group and control group) will be studied by upper endoscopy with Magniview™ scopes and EPK-i7010 processor (OE system™).

The technique involves the use of a distal rubber hood (OE-A58) at the tip of the scope (EG-2990Zi). After reaching the line Z, the four quadrants of the three levels of the esophagus (upper, middle and lower esophagus) will be evaluated in the same way. The cup will contact to the esophageal mucosa and water will be instilled. Initially only the OE system™ will be used (mode 1) If there is no evidence of minimal changes, the optical magnification will be implemented through the actions of a button on the Magniview scope. Finally the OE system™ will be off and only the Magniview™ will be used with white light.

All changes seen will be recorded (by video and pictures) in the specific phase of the study (OE system™ alone, OE system™ with Magniview™ or Magniview™ alone). Finally, biopsies will be taken in both groups (one of each esophagus level randomly and one targeted biopsy to any lesion). The endoscopies will be performed by three endoscopist blind to the group selection and trained on this new technology (all of them with more than 10 procedures).

Mucosal minimal changes will be evaluated as the Sharma et al. classification:

1. IPCLs (number, dilatation, and tortuosity). Dilatation of IPCLs will be recognized as a change in the pattern characterized by increased size or caliber of individual IPCLs. Tortuosity is define by the presence of corkscrewing or the twisted nature of individual IPCLs.
2. Presence of microerosions (definitive mucosal breaks not visible at standard endoscopy).
3. Vascularity at the squamocolumnar junction.
4. Presence of columnar island in the distal esophagus.
5. Ridge-villous pattern below the squamocolumnar junction characterized by the presence of uniform, longitudinally aligned ridges alternating with a villiform pattern.

Interobserver and Intraobserver Agreement: A data set containing pictures of the three esophagus levels in the three phase of the study (OE system™ alone, OE system™ with Magniview™ or Magniview™ alone) will be presented to three blinded endoscopists, who will confirm or not the findings. Inter- and intraobserver reproducibility will be measured based on comparison of still images between the three investigators. To evaluate the intraobserver agreement each investigator will assess the images three times and the answers will be compared. To evaluate the interobserver agreement all answers between the three investigators will be compared.

Statistical analysis: Baseline characteristics as age, gender, body mass index, symptoms will be compared between case and control group using Chi-square o Fisher Test for categorical variable, and for continuing variables, we will use the Mann-Whitney Test. Diagnosis efficacy will be measured thought sensitive, specificity and accuracy. All the statistical analysis will be performed using SPSS software suite v.22.

Limitations

* Only patients with typical reflux symptoms will participate in the study (heartburn or regurgitation).
* The protocol will be performed in only one center.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old patients
* Who agree to participate in the study
* Patients with reflux symptoms (heartburn and regurgitation), with8 or more points at the GERD questionnaire and no evidence of ulcerative esophagitis, esophageal strictures, Barrett's esophagus or any erosive sign according to Los Angeles classification (Grade A to D) in the upper endoscopy using white light nor I-Scan™

Exclusion Criteria:

* Patients with ulcerative esophagitis, esophageal strictures, Barrett's esophagus or any erosive sign according to Los Angeles classification (Grade A to D)
* Patients with medical history of any kind of esophagitis (including actinic, caustic or eosinophilic), achalasia.
* Esophageal varices
* Patients with evidence of cancer or mass lesion in the esophagus
* Protons bump inhibitor consumption for at least 3 weeks before endoscopy
* Inability to discontinue non steroidal anti-inflammatory drugs or aspirin prior to the study
* Severe uncontrolled coagulopathy
* Gastric lesions (ulcer, polyp, cancer), severe gastroparesis
* Prior history of esophageal or gastric surgery.
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that had reflux symptoms (heartburn and regurgitation) and 8 or more points at the Spanish version of GERD questionnaire validated by Zavala-González et al. underwent an upper videoendoscopy using initially high definition white light and then digital chromoendoscopy (I-Scan™) in the three different image algorithms. If the esophagus was normal and no changes were seen by these two techniques, they were considered as NERD patients and a pH-impedanciometry was performed as gold standard study, in order to diagnosis reflux disease. We considered a GERD diagnosis with more than 73 episodes of reflux in 24 hours or acid exposure time abnormal with ph<4 measured in more than 4,2%of the time over 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Digital chromoendoscopy and optical magnification in the diagnosis of intrapapillary loops (IPCLs) in esophagus. Number of participants with increased number of IPCLs, dilatation or tortuosity of IPCLs | two months

SECONDARY OUTCOMES:
Number of patients in whom the minimal esophageal changes are diagnosed by the digital chromoendoscopy without using the magnification, or with the magnification without using the digital chromoendoscopy or using both. | two months
Number of patients with increased number, dilatation or tortuosity of the intrapapilary loops on endoscopic image and have a positive biopsy for inflammation of mucosa. | two months

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Robles-Medranda, MD, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Omnihospital, Guayaquil, Guayas, Ecuador

REFERENCES:
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Kasap E, Zeybel M, Asik G, Ayhan S, Yuceyar H. Correlation among standard endoscopy, narrow band imaging, and histopathological findings in the diagnosis of nonerosive reflux disease. J Gastrointestin Liver Dis. 2011 Jun;20(2):127-30. PMID 21725507
- [Background] Zentilin P, Savarino V, Mastracci L, Spaggiari P, Dulbecco P, Ceppa P, Savarino E, Parodi A, Mansi C, Fiocca R. Reassessment of the diagnostic value of histology in patients with GERD, using multiple biopsy sites and an appropriate control group. Am J Gastroenterol. 2005 Oct;100(10):2299-306. doi: 10.1111/j.1572-0241.2005.50209.x. PMID 16181384
- [Background] Kim MS, Choi SR, Roh MH, Lee JH, Jang JS, Kim BG, Kim SO, Han JS, Hsing CT. Efficacy of I-scan endoscopy in the diagnosis of gastroesophageal reflux disease with minimal change. Clin Endosc. 2011 Sep;44(1):27-32. doi: 10.5946/ce.2011.44.1.27. Epub 2011 Sep 30. PMID 22741109
- [Background] Zavala-Gonzales MA, Azamar-Jacome AA, Meixueiro-Daza A, Ramos A, J JR, Roesch-Dietlen F, Remes-Troche JM. Validation and diagnostic usefulness of gastroesophageal reflux disease questionnaire in a primary care level in Mexico. J Neurogastroenterol Motil. 2014 Oct 30;20(4):475-82. doi: 10.5056/jnm14014. PMID 25273118
- [Background] Kandulski A, Weigt J, Caro C, Jechorek D, Wex T, Malfertheiner P. Esophageal intraluminal baseline impedance differentiates gastroesophageal reflux disease from functional heartburn. Clin Gastroenterol Hepatol. 2015 Jun;13(6):1075-81. doi: 10.1016/j.cgh.2014.11.033. Epub 2014 Dec 9. PMID 25496815
- [Background] Dent J, Armstrong D, Delaney B, Moayyedi P, Talley NJ, Vakil N. Symptom evaluation in reflux disease: workshop background, processes, terminology, recommendations, and discussion outputs. Gut. 2004 May;53 Suppl 4(Suppl 4):iv1-24. doi: 10.1136/gut.2003.034272. PMID 15082609
- [Background] Sharma P, Wani S, Bansal A, Hall S, Puli S, Mathur S, Rastogi A. A feasibility trial of narrow band imaging endoscopy in patients with gastroesophageal reflux disease. Gastroenterology. 2007 Aug;133(2):454-64; quiz 674. doi: 10.1053/j.gastro.2007.06.006. Epub 2007 Jun 8. PMID 17681166
- [Background] Kumagai Y, Toi M, Inoue H. Dynamism of tumour vasculature in the early phase of cancer progression: outcomes from oesophageal cancer research. Lancet Oncol. 2002 Oct;3(10):604-10. doi: 10.1016/s1470-2045(02)00874-4. PMID 12372722
- [Background] Lundell LR, Dent J, Bennett JR, Blum AL, Armstrong D, Galmiche JP, Johnson F, Hongo M, Richter JE, Spechler SJ, Tytgat GN, Wallin L. Endoscopic assessment of oesophagitis: clinical and functional correlates and further validation of the Los Angeles classification. Gut. 1999 Aug;45(2):172-80. doi: 10.1136/gut.45.2.172. PMID 10403727
- [Background] Neumann H, Fujishiro M, Wilcox CM, Monkemuller K. Present and future perspectives of virtual chromoendoscopy with i-scan and optical enhancement technology. Dig Endosc. 2014 Jan;26 Suppl 1:43-51. doi: 10.1111/den.12190. Epub 2013 Oct 23. PMID 24373000
- [Result] Gomes CA Jr, Loucao TS, Carpi G, Catapani WR. A study on the diagnosis of minimal endoscopic lesions in nonerosive reflux esophagitis using computed virtual chromoendoscopy (FICE). Arq Gastroenterol. 2011 Jul-Sep;48(3):167-70. doi: 10.1590/s0004-28032011000300002. PMID 21952699